CLINICAL TRIAL: NCT02121444
Title: BETAEVAL - The New BETACONNECT® Auto-injector: Adherence and EVALuation of MS Patients Treated With Betaferon®
Brief Title: BAY86-5046 (Betaseron), Non Interventional Studies
Acronym: BETAEVAL
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17101; BF1414DE (Other: Company internal)
Record Dates: First submitted 2014-04-22; First posted 2014-04-23 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Multiple Sclerosis
Keywords: RRMS; CIS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Multiple Sclerosis patients who are treated with Betaferon and who are using the Betaconnect auto-injector
  Interventions: Drug: Interferon beta-1b (Betaferon, BAY 86-5046); Device: BETACONNECT auto-injector.

INTERVENTIONS:
Drug: Interferon beta-1b (Betaferon, BAY 86-5046)
Device: BETACONNECT auto-injector.

SUMMARY:
This study aims to investigate adherence to therapy among patients treated with Betaferon who are using the BETACONNECT autoinjector.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of relapsing remitting multiple sclerosis or a clinically isolated syndrome.
* Patients must be on treatment with Betaferon or the decision to treat patients with Betaferon has been made by the attending physician.
* Patient and attending physicians must have agreed on the usage of the BETACONNECT auto-injector device
* Written informed consent must be obtained.

Exclusion Criteria:

* Patients receiving any other disease modifying drug.
* Contraindications of Betaferon described in the Summary of Product Characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with relapsing remitting multiple sclerosis (RRMS) or patients with a clinically isolated syndrome (CIS) who are treated with Betaferon or will be treated with Betaferon according to the attending physician's decision and for whom the patient and the physician have agreed to use the BETACONNECT device.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2016-03-09 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Adherence measure to Betaferon therapy based on the real BETACONNECT injections | up to 24 weeks
  Adherence to therapy will be defined as applying ≥80% of prescribed Betaferon dosages, which can be derived from electronic data stored in the BETACONNECT device.

SECONDARY OUTCOMES:
Satisfaction with and evaluation of the BETACONNECT auto-injector recorded by patient questionnaire | up to 24 weeks
Evaluation of health related quality of life,measured with the self-administered Functional Assessment of Multiple Sclerosis (FAMS) questionnaire | up to 24 weeks
Evaluation of Anxiety measured with the self-administered Hospital Anxiety and Depression Scale (HADS) | up to 24 weeks
Evaluation of Depression measured with the self-administered Center for Epidemiologic Studies Depression Scale (CES-D) | up to 24 weeks
Evaluation of Fatigue measured with the self-administered Fatigue Scale for Motor and Cognitive functions (FSMC) | up to 24 weeks
Evaluation of Cognition will be measured by the HCP with the Symbol Digit Modalities Test (SDMT) | up to 24 weeks
Local skin reactions recorded by Health Care Provider (HCP) evaluation | up to 24 weeks
Evaluation of injection-related specifics such as injection date, time, and speed will be recorded by the BETACONNECT device | up to 24 weeks
Number of Treatment-emergent Adverse Events (TEAE) | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Germany

REFERENCES:
- [Derived] Kleiter I, Lang M, Jeske J, Norenberg C, Stollfuss B, Schurks M. Adherence, satisfaction and functional health status among patients with multiple sclerosis using the BETACONNECT(R) autoinjector: a prospective observational cohort study. BMC Neurol. 2017 Sep 6;17(1):174. doi: 10.1186/s12883-017-0953-8. PMID 28877664